CLINICAL TRIAL: NCT00160225
Title: A Randomized, Double-Blind, Placebo Controlled, Two-Treatment and Two-Period Cross-Over, Mono-Center Study to Evaluate the Efficacy and Safety of Daglutril 300 mg Once Daily Compared to Placebo on Top of Losartan in Type 2 Diabetics With Overt Nephropathy and Well Controlled Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of Daglutril Compared to Placebo on Top of Losartan in Type 2 Diabetics With Overt Nephropathy and Well Controlled Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S306.2.009; 2004-001980-24
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
Keywords: blood pressure, diabetic nephropathy, proteinuria
MeSH Terms: conditions — Hypertension; Diabetic Nephropathies; Proteinuria | interventions — SLV 306

INTERVENTIONS:
Drug: Daglutril

SUMMARY:
This study is to evaluate the end of treatment effect of Daglutril compared to placebo on top of losartan.

ELIGIBILITY:
Inclusion Criteria:

* treated with optimized dose of losartan (constant dose for at least four weeks before randomization and throughout the whole study period) for at least four weeks
* urinary albumin excretion ≥ 20 and < 1000 µg/min
* sitting systolic/diastolic blood pressure (SBP/DBP) < 140/90 mmHg at the end of placebo run-in phase

Exclusion Criteria:

* known secondary hypertension
* decompensated congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Ranica, Italy

REFERENCES:
- [Derived] Parvanova A, van der Meer IM, Iliev I, Perna A, Gaspari F, Trevisan R, Bossi A, Remuzzi G, Benigni A, Ruggenenti P; Daglutril in Diabetic Nephropathy Study Group. Effect on blood pressure of combined inhibition of endothelin-converting enzyme and neutral endopeptidase with daglutril in patients with type 2 diabetes who have albuminuria: a randomised, crossover, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2013 Sep;1(1):19-27. doi: 10.1016/S2213-8587(13)70029-9. Epub 2013 Jun 13. PMID 24622263